CLINICAL TRIAL: NCT07266857
Title: Pilot Observational Comparative Study Evaluating the Impact of the e-Bug Educational Programme on Parental Consent and HPV Vaccination Coverage During the National School-Based Vaccination Campaign in a Middle School in the Alpes-Maritimes
Brief Title: Impact of an e-Bug Educational Intervention on HPV Vaccine Uptake in Middle School Students
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25SantéMentale02
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Papillomavirus Infection; Papillomavirus Vaccines; Vaccination Coveage
MeSH Terms: conditions — Papillomavirus Infections | interventions — Consent Forms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot School Using e-Bug Programme
  Interventions: Other: Consent for HPV vaccination
- Other Middle Schools in Alpes-Maritimes Department
  Interventions: Other: Consent for HPV vaccination

INTERVENTIONS:
Other: Consent for HPV vaccination — Consent for HPV vaccination

SUMMARY:
This study is a non-interventional observational pilot analysis assessing the possible impact of an educational programme (e-Bug) on parental consent and HPV vaccination uptake during the 2023-2024 and 2024-2025 national school-based HPV vaccination campaigns in France. The study focuses on one middle school in the Alpes-Maritimes department where teachers and the school nurse had been previously trained on HPV and used e-Bug educational resources in class as part of routine health education. No research-related intervention was conducted, and the educational programme was not introduced or modified for the purpose of the study. Only aggregated and anonymised vaccination data were used. These data were routinely collected by the Regional Health Agency (ARS PACA) as part of the national vaccination programme and transmitted for analysis. Aggregated data from the pilot school were compared with departmental-level outcomes to describe whether an upstream educational approach may be associated with improved parental acceptance and higher HPV vaccination coverage. This study aims to contribute to the understanding of educational determinants of vaccine uptake in a real-life school setting without involving any participant recruitment or individual data collection.

ELIGIBILITY:
Inclusion Criteria:

* No individual participants are enrolled. The study uses only aggregated, anonymised vaccination data routinely collected by ARS PACA

Exclusion Criteria:

* Not applicable. No individual-level inclusion or exclusion criteria are defined, as no participants are enrolled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Aggregated data from 5th-grade students enrolled in one pilot middle school using the e-Bug programme, compared with aggregated data from all other middle schools in the Alpes-Maritimes department. No individual-level data were accessed.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination uptake (1st and 2nd doses) in the pilot school compared with departmental data | From (start of 2023-2024 HPV vaccination campaign) to(end of 2024-2025)
  e-Bug educational programme

SECONDARY OUTCOMES:
Parental consent rate (acceptability) | From (start of 2023-2024 HPV vaccination campaign) to(end of 2024-2025)
  Aggregated proportion of parents providing positive consent for HPV vaccination in the pilot school, compared with aggregated departmental consent rates collected by ARS PACA during the 2023-2024 and 2024-2025 school-based campaigns.
Response rate (return of vaccination authorisation forms) | From (start of 2023-2024 HPV vaccination campaign) to(end of 2024-2025)
  Aggregated rate of returned parental authorisation forms (regardless of response: yes/no) in the pilot school compared with departmental response rates.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France